CLINICAL TRIAL: NCT07357948
Title: Omission of Surgery for Triple-negative Breast Cancer in Complete Response Confirmed by MRI and Macrobiopsy After Neoadjuvant Chemo-immunotherapy: a Randomized, Multicenter Phase II Trial.
Brief Title: Omission of Surgery for Triple-negative Breast Cancer in Complete Response After Neoadjuvant Chemo-immunotherapy
Acronym: WISH-OMICHIR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IC 2025-05; 2025-A02926-43 (Other: ANSM)
Record Dates: First submitted 2026-01-05; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Triple Negative Breast Cancer; Non-Metastatic
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): standard care, except surgery
  Interventions: Procedure: Omission of surgery
- Control (No Intervention): standard care, including surgery

INTERVENTIONS:
Procedure: Omission of surgery — Patients will not undergo breast and axillary surgery.
  Arms: Experimental

SUMMARY:
This clinical study aims to determine if skipping breast and axillary surgery could provide similar control of local and distant disease, with fewer complications and better quality of life, for triple-negative breast cancer patients in complete response after neoadjuvant chemo-immunotherapy.

Patients will be randomised into 2 groups :

* Control arm will receive the standard treatment, including surgery
* Experimental arm will receive the standard treatment, except surgery

ELIGIBILITY:
Inclusion Criteria:

1. Sex and age: Female, aged 18 years or older.
2. Histological type: Invasive breast carcinoma of no special type (NST).
3. Triple-negative phenotype, defined by:

   * Estrogen receptor (ER) < 10%,
   * Progesterone receptor (PR) < 10%,
   * HER2-negative status according to ASCO/CAP criteria (IHC score 0-1+, or 2+ without amplification by in situ hybridization).
4. High proliferation index: Ki-67 > 30%.
5. Primary tumor classified as T2, i.e. tumor size between 2 and 5 cm on imaging at diagnosis (mammography, ultrasound, and breast MRI).
6. No regional lymph node involvement or distant metastasis, confirmed by 18F-FDG PET-CT performed prior to neoadjuvant treatment.
7. Completion of the full neoadjuvant chemo-immunotherapy (NCIT) protocol according to the KEYNOTE-522 regimen (≥7 cycles including pembrolizumab).
8. Breast-conserving surgery deemed feasible based on the initial surgical assessment.
9. Radiological complete response (rCR) on post-NCIT breast MRI, associated with a negative vacuum-assisted biopsy (VAB) of the clip-marked tumor bed, confirming the absence of residual invasive or in situ disease.
10. Written informed consent obtained prior to any study-specific procedure.
11. Ability of the patient to comply with the protocol requirements and scheduled follow-up.
12. Affiliation with a national health insurance system, in accordance with French regulations.

Exclusion Criteria:

1. Presence of regional recurrence or metastatic disease at inclusion.
2. History of thoracic, breast, or regional lymph node irradiation, regardless of indication.
3. Invasive lobular carcinoma, excluded due to its different response profile and increased risk of multifocal residual disease.
4. Presence of ductal carcinoma in situ (DCIS) on diagnostic biopsy, or diffuse suspicious microcalcifications on mammography, precluding reliable assessment of complete response.
5. Bilateral breast cancer (except for localized and treated contralateral DCIS), or history of ipsilateral or contralateral invasive breast cancer.
6. Multifocal or multicentric disease detected on imaging (mammography, ultrasound, or breast MRI).
7. Skin involvement or inflammatory breast cancer, identified on imaging or clinical examination.
8. History of malignancy other than breast cancer, unless the disease has been in complete remission for ≥ 5 years and is considered at low risk of recurrence, with the exception of:

   * Treated carcinoma in situ of the cervix, endometrium, or colon,
   * Melanoma in situ,
   * Completely excised cutaneous basal cell or squamous cell carcinoma.
9. Severe or progressive non-malignant disease limiting life expectancy to less than 10 years, in the investigator's judgment.
10. Presence of a high-risk germline mutation predisposing to breast cancer (including BRCA1, BRCA2, or other identified predisposition genes).
11. Participation in another interventional clinical trial within 30 days prior to inclusion.
12. Current pregnancy or breastfeeding.
13. Cognitive impairment, psychiatric disorder, or social situation preventing valid informed consent or adequate understanding of the protocol, as assessed by the investigator.
14. Individuals deprived of liberty or under legal protection (guardianship, curatorship, or similar legal status), in accordance with applicable regulations.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-08-01 (Estimated); Primary Completion 2031-07-31 (Estimated); Study Completion 2033-07-31 (Estimated)

PRIMARY OUTCOMES:
Assess invasive disease-free survival (iDFS) | Within 36 months after randomisation
  Disease-free survival rate, taking into account the first occurrence of any of the following events : local or regional invasive recurrence, contralateral invasive breast cancer, distant metastasis, second primary cancer, death from any cause.

SECONDARY OUTCOMES:
Assessing the locoregional recurrence-free interval (LRFI) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Number of months between randomization and the first occurrence of local or regional invasive recurrence (in the breast or regional lymph nodes)
Assessing distant recurrence-free interval (DRFI) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Number of months between randomization and the first occurrence of distant metastases
Assessing overall survival (OS) | From date of randomisation until the date of death, assessed up to 60 months
  Number of months between randomization and death, regardless of cause
Assessing the adverse effects of macrobiopsy | Up to 30 days after macrobiopsy
  Number of adverse events
Assessing the adverse effects of standard of care radiotherapy treatment | From start of treatment through study completion, an average of 60 months
  Number of grade ≥ 3 adverse events related to radiotherapy
Assessing quality of life - EORTC QLQ-C30 Physical Functioning score | Randomisation, month 6, month 12, month 18, month 24, month 30, month 36
  EORTC QLQ-C30 Physical Functioning score (0-100; higher = better)
Assessing quality of life - EORTC QLQ-C30 Fatigue score | Randomisation, month 6, month 12, month 18, month 24, month 30, month 36
  EORTC QLQ-C30 Fatigue score (0-100; higher = worse)
Assessing quality of life - EORTC QLQ-C30 Global Health Status/Quality of Life score | Randomisation, month 6, month 12, month 18, month 24, month 30, month 36
  EORTC QLQ-C30 Global Health Status/Quality of Life score (0-100; higher = better)
Assessing quality of life and aesthetic results - EORTC QLQ-BR42 Body Image score | Randomisation, month 6, month 12, month 18, month 24, month 30, month 36
  EORTC QLQ-BR42 Body Image score (0-100; higher = better)
Assessing quality of life and aesthetic results - EORTC QLQ-BR42 Arm Symptoms score | Randomisation, month 6, month 12, month 18, month 24, month 30, month 36
  EORTC QLQ-BR42 Arm Symptoms score (0-100; higher = worse)
Assessing quality of life and aesthetic results - EORTC QLQ-BR42 Future Perspective score | Randomisation, month 6, month 12, month 18, month 24, month 30, month 36
  EORTC QLQ-BR42 Future Perspective score (0-100; higher = better)
Assessing the number of benign biopsies during follow-up | From date of randomisation until the date of new biopsy, assessed up to 60 months
  Number of benign biopsies of the breast or ipsilateral lymph nodes performed during follow-up
Number of patients with residual disease not detected in the control arm | At surgery
  Evaluating the performance of MRI and macrobiopsy for predicting complete histologic response (pCR)

CONTACTS AND LOCATIONS:
Overall Officials: Toulsie Ramtohul, MD, Principal Investigator — Institut Curie

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months
Access Criteria: ccess to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).